CLINICAL TRIAL: NCT03691831
Title: A Phase 3 Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study of A-101 Topical Solution Applied Twice a Week in Subjects With Common Warts
Brief Title: A Study of A-101 Topical Solution for the Treatment of Common Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-101-WART-302
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Common Wart
MeSH Terms: conditions — Warts | interventions — Exercise; 2-Propanol

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded vehicle solution is packaged to match the active study drug and will be stored under the same conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): A-101 45% (Topical solution, hydrogen peroxide 45%)
  Interventions: Drug: Active
- Vehicle (Placebo Comparator): Topical solution, isopropyl alcohol and water
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Active — A-101 45% (hydrogen peroxide 45% topical solution)
  Other Names: hydrogen peroxide 45%
  Arms: Active
Other: Vehicle — Vehicle solution containing isopropyl alcohol and water
  Other Names: isopropyl alcohol and sterile water
  Arms: Vehicle

SUMMARY:
Phase 3 Study of A-101 Topical Solution in Subjects with Common Warts

DETAILED DESCRIPTION:
A Phase 3 Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of A-101 Topical Solution Applied Twice a Week in Subjects with Common Warts

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal guardian is able to comprehend and is willing to sign an informed consent/assent for participation in this study.
2. Male or female ≥ 2 years old.
3. Subject has a clinical diagnosis of common warts (verruca vulgaris).
4. Subject has at least 1 and up to 6 clearly identifiable common warts located on the trunk or extremities that meet the requirements as defined below:

   1. Have a longest axis that is ≥3 and ≤8 mm and have a thickness of ≤3mm
   2. Be a discrete lesion, i.e. each wart meeting the entry criteria is clearly separated from other warts.
   3. Be present for at least 4 weeks
   4. Not be covered with hair which, in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   5. Not be in an intertriginous fold
   6. Periungual, subungual, genital, anal, mosaic, plantar, flat and filiform warts are excluded from treatment and evaluation. If a subject has these types of warts, but also has warts that meet the inclusion criteria, the subject will NOT be excluded from the study.
5. Each common wart identified for treatment must have a PWA ≥ 2.
6. Subject's chemistry and complete blood count results are within normal limits. If any of the laboratory values are outside normal range, the treating investigator must assess the value(s) as NOT clinically significant and document this in the subject's medical chart in order for the subject to be eligible for randomization.
7. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair the evaluation of the identified common warts or which exposes the subject to an unacceptable risk by study participation.
8. Subject is willing and able to follow all study instructions and to attend all study visits.
9. Subject must be the only individual in a household participating in the study.

Exclusion Criteria:

1. Subject has clinically atypical common warts.
2. Subject is immunocompromised (e.g., due to chemotherapy, systemic steroids, genetic immunodeficiency, transplant status, etc.).
3. Subject has a history of Human Immunodeficiency Virus (HIV) infection.
4. Subject has had any Human Papilloma Virus (HPV) vaccine within 6 months prior to Visit 1.
5. Subject has used any of the following intralesional therapies within the specified period prior to Visit 2:

   1. Immunotherapy (e.g., Candida antigen, mumps antigen, Trichophyton antigen); 8 weeks
   2. Anti-metabolite therapy (e.g., bleomycin, 5-fluorouracil); 8 weeks
6. Subject has used any of the following systemic therapies within the specified period prior to Visit 2:

   1. Immunomodulatory/immunosuppressant therapy (e.g., etanercept, alefacept, infliximab); 16 weeks
   2. Glucocorticosteroids (inhaled and intra-nasal steroids are permitted); 28 days
7. Subject has used any of the following topical therapies within the specified period prior to Visit 2 on, or in the proximity to any of the common warts identified for treatment, that in the investigator's opinion interferes with the study medication treatment or the study assessments:

   1. LASER, light or other energy-based therapy (e.g., intense pulsed light [IPL], photodynamic therapy [PDT]); 180 days
   2. Immunotherapy (e.g., imiquimod, squaric acid dibutyl ester[SADBE], etc.) 12 weeks
   3. Liquid nitrogen, electrodesiccation, curettage; 60 days
   4. Hydrogen peroxide; 90 days
   5. Antimetabolite therapy (e.g., 5-fluorouracil); 8 weeks
   6. Retinoids; 90 days
   7. Over-the-counter (OTC) wart therapies and cantharidin; 28 days
8. Subject currently has or has had any of the following within the specified period prior to Visit 1 on or in the proximity to any of the common warts identified for treatment that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

   1. Cutaneous malignancy; 180 days
   2. Sunburn; currently
   3. Pre-malignancy (e.g., actinic keratosis); currently
9. Subject has a history of sensitivity to any of the ingredients in the study medications.
10. Subject has any current skin or systemic disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
11. Participation in another therapeutic investigational drug/device trial in which administration of an investigational treatment occurred with 30 days prior to Visit 1.
12. Subject has an active malignancy.
13. Subjects is viewed by the Principal Investigator as not being able to complete the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Schynder, Study Director — Aclaris Therapeutics
Locations (24):
- United States (24):
  - Aclaris Investigational Site, Glendale, Arizona
  - Aclaris Investigational Site, Fort Smith, Arkansas
  - Aclaris Investigational Site, Encinitas, California
  - Aclaris Investigational Site, San Diego, California
  - Aclaris Investigational Site, Denver, Colorado
  - Aclaris Investigational Site, Coral Gables, Florida
  - Aclaris Investigational Site, Miami, Florida
  - Aclaris Investigational Site, New Albany, Indiana
  - Aclaris Investigational Site, Rockville, Maryland
  - Aclaris Investigational Site, Quincy, Massachusetts
  - Aclaris Investigational Site, Saint Joseph, Missouri
  - Aclaris Investigational Site, Omaha, Nebraska
  - Aclaris Investigational Site, Rochester, New York
  - Aclaris Investigational Site, Raleigh, North Carolina
  - Aclaris Investigational Site, Beachwood, Ohio
  - Aclaris Investigational Site, Upper Saint Clair, Pennsylvania
  - Aclaris Investigational Site, Anderson, South Carolina
  - Aclaris Investigational Site, Knoxville, Tennessee
  - Aclaris Investigational Site, Nashville, Tennessee
  - Aclaris Investigational Site, Arlington, Texas
  - Aclaris Investigational Site, College Station, Texas
  - Aclaris Investigational Site, Houston, Texas
  - Aclaris Investigational Site, Lynchburg, Virginia
  - Aclaris Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Topical solution, hydrogen peroxide 45%
  A-101: hydrogen peroxide 45% topical solution
Period: Overall Study
Arm/Group | Active | Vehicle
Started | 251 | 251
Completed | 224 | 220
Not Completed | 27 | 31
Not completed — Lost to Follow-up | 16 | 12
Not completed — Withdrawal by Subject | 9 | 17
Not completed — Investigator Decision | 2 | 2

BASELINE CHARACTERISTICS:
Population: randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Vehicle | Total
Number analyzed (Participants) | 251 | 251 | 502
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 70 | 145
  Between 18 and 65 years | 169 | 168 | 337
  >=65 years | 7 | 13 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (17.80) | 31.7 (17.33) | 31.4 (17.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 111 | 215
  Male | 147 | 140 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 35 | 58
  Not Hispanic or Latino | 206 | 199 | 405
  Unknown or Not Reported | 22 | 17 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 13 | 13 | 26
  White | 228 | 230 | 458
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 251 | 251 | 502
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 9 | 14 | 23
  II - Burns Easily | 93 | 91 | 184
  III - Burns Moderately | 87 | 83 | 170
  IV - Burns Minimally | 42 | 41 | 83
  V - Rarely Burns | 13 | 14 | 27
  VI - Never Burns | 7 | 8 | 15
Prior Treatment of any Wart Treated [Count of Participants; unit: Participants]
  Yes | 114 | 112 | 226
  No | 137 | 139 | 276
Total Warts Treated [Count of Participants; unit: Participants]
  1 | 126 | 142 | 268
  2 | 68 | 49 | 117
  3 | 22 | 18 | 40
  4 | 13 | 14 | 27
  5 | 10 | 10 | 20
  6 | 12 | 18 | 30
Time Since First Appearance of Most Recent Wart Treated [Mean (Standard Deviation); unit: days] | 1726.7 (2210.95) | 1670.2 (2041.81) | 1698.6 (2126.62)
Time since First Appearance of Least Recent Wart Treated [Mean (Standard Deviation); unit: days] | 1926.2 (2298.39) | 1780.0 (2037.01) | 1853.5 (2171.47)
Thickness of "Largest" Wart Treated [Mean (Standard Deviation); unit: millimeters] | 1.49 (0.741) | 1.50 (0.752) | 1.49 (0.746)
Longest Axis of "Largest" Wart Treated [Mean (Standard Deviation); unit: millimeter] | 5.1 (1.54) | 5.1 (1.55) | 5.1 (1.55)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is the Number of Subjects Whose Identified Common Warts Are Determined to be Clear on the PWA Scale (PWA=0) at Visit 10 (Day 60)
Description: The primary efficacy endpoint is the number of subjects whose identified common warts are determined to be clear on the Physician Wart Assessment (PWA) scale (PWA=0) at Visit 10 (Day 60).
  Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 60
Population: The study's primary endpoint was to evaluate the amount of patients achieving a clearance of all baseline WARTS. Patients were stratified by the amount of WARTS at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 251 | 251
Participants
  Warts at Baseline - All | 33 | 8
  Warts at Baseline - 1: number analyzed (Participants) | 126 | 142
  Warts at Baseline - 1 | 19 | 4
  Warts at Baseline - 2: number analyzed (Participants) | 68 | 49
  Warts at Baseline - 2 | 9 | 0
  Warts at Baseline - 3: number analyzed (Participants) | 22 | 18
  Warts at Baseline - 3 | 3 | 0
  Warts at Baseline - >3: number analyzed (Participants) | 35 | 42
  Warts at Baseline - >3 | 2 | 4
Statistical Analysis 1: Comparison: Active vs Vehicle; A summary of the wart clearance at Visit 10; Test type: Superiority; p = 0.0001, Mixed Models Analysis — P-Value test comparing the Patients Cleared of All Baseline Warts in the Active (A-101 45%) and vehicle groups; Odds Ratio (OR) = 4.80, 95% CI 2-sided [2.14 to 10.76]

2. Secondary Outcome: Number of Subjects With Complete Clearance of All Treated Common Warts Between Active and Vehicle on the Physician Wart Assessment (PWA) Scale (PWA=0) at Visit 13 (Day 137)
Description: Number of subjects whose identified common warts are determined to be clear on the Physician Wart Assessment (PWA) scale (PWA=0) at Visit 13 (Day 137).
  Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 137
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 251 | 251
Participants
  Warts at Baseline - All | 56 | 25
  Warts at Baseline - 1: number analyzed (Participants) | 126 | 142
  Warts at Baseline - 1 | 29 | 13
  Warts at Baseline - 2: number analyzed (Participants) | 68 | 49
  Warts at Baseline - 2 | 12 | 2
  Warts at Baseline - 3: number analyzed (Participants) | 22 | 18
  Warts at Baseline - 3 | 5 | 2
  Warts at Baseline - >3: number analyzed (Participants) | 35 | 42
  Warts at Baseline - >3 | 10 | 8
Statistical Analysis 1: Comparison: Active vs Vehicle; P-Value test comparing the Patients Cleared of All Baseline Warts in the Active (A-101 45%) and vehicle groups; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.71, 95% CI 2-sided [1.61 to 4.56]

3. Secondary Outcome: Mean Per-Subject Percent of All Warts That Were Clear on the Physician Wart Assessment (PWA) Scale Between Active and Vehicle That Are Clear (PWA=0) at Visit 13 (Day 137)
Description: Mean Per-Subject Percent of all Warts that were Clear on the Physician Wart Assessment (PWA) scale between Active (A-101 45%) and Vehicle that are clear (PWA=0) at Day 137.
  Clearance of all treated warts will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 137
Measure: Mean (Standard Deviation); unit: percentage of warts cleared
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 251 | 251
percentage of warts cleared | 27.7 (2.30) | 12.2 (2.30)
Statistical Analysis 1: Comparison: Active vs Vehicle; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 15.44, 95% CI 2-sided [9.0 to 21.8]

4. Secondary Outcome: Number of Subjects With a Single Wart at Baseline Whose Wart Was Clear on the PWA Scale Between Active and Vehicle Group (PWA=0) at Visit 10 (Day 60)
Description: Comparison between Active (A-101 45%) and Vehicle of subjects with a single wart at baseline, whose wart is clear (PWA=0) at Day 60.
  Clearance of the single wart at baseline will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 126 | 142
Participants | 19 | 4
Statistical Analysis 1: Comparison: Active vs Vehicle; Test type: Superiority; p = 0.0006, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 5.20, 95% CI 2-sided [1.76 to 15.53]

5. Secondary Outcome: Median Time for Subjects to Achieve Clearance (PWA=0) of All Treated Common Warts
Description: Comparison between Active (A-101 45%) and Vehicle with respect to the median time to achieve onset of clearance (PWA=0) for all treated warts at Day 137.
  Clearance of all treated warts will be assessed using the Physician Wart Assessment (PWA) scale which is a four point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Day 137
Population: A median was not able to be calculated in the Vehicle group due to an insufficient number of participants with events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 251 | 251
days | 113 [79.0 to 114.0] | NA [NA to NA] — A median was not able to be calculated in the Vehicle group due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Active vs Vehicle; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 3.33

ADVERSE EVENTS:
Time Frame: 137 days; Treatment-emergent adverse events (TEAEs) had a start date on or after the date of Visit 2 (study day 1) and treatment-emergent serious adverse events had a start date on or after the date of Visit 1 (Screening). Collection continued through visit 11 (Day 78)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Arm/Group | Active | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/251
Serious Adverse Events (participants affected / at risk) | 1/251 | 2/251
Other Adverse Events (participants affected / at risk) | 154/251 | 61/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=251) | Vehicle (N=251)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — The event onset was 50 days after the last study treatment application, therefore not treatment-emergent
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=251) | Vehicle (N=251)
Vomiting (Gastrointestinal disorders) | 1 | 2
Application site dermatitis (General disorders) | 3 | 1
Application site discoloration (General disorders) | 4 | 1
Application site dryness (General disorders) | 2 | 0
Application site erosion (General disorders) | 13 | 4
Application site erythema (General disorders) | 26 | 10
Application site irritation (General disorders) | 5 | 0
Application site edema (General disorders) | 10 | 5
Application site pain (General disorders) | 107 | 5
Application site pallor (General disorders) | 44 | 0
Application site paresthesia (General disorders) | 3 | 3
Application site pruritus (General disorders) | 23 | 3
Application site scab (General disorders) | 20 | 1
Nasopharyngitis (Infections and infestations) | 7 | 3
Sinusitis (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 11 | 6
Influenza (Infections and infestations) | 2 | 5
Pharyngitis streptococcal (Infections and infestations) | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Application site haemorrhage (General disorders) | 1 | 0
Application site hypoaesthesia (General disorders) | 1 | 0
Application site swelling (General disorders) | 1 | 0
Application site ulcer (General disorders) | 1 | 0
Application site vesicles (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Bronchitis (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Ear Infection (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Face Injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03691831/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03691831/SAP_002.pdf
  • Informed Consent Form (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03691831/ICF_006.pdf